CLINICAL TRIAL: NCT06594640
Title: A Multicenter, Prospective Phase I/II Trial to Evaluate the Safety and Efficacy of Mitoxantrone Hydrochloride Liposome in Combination With Cyclophosphamide, Vincristine, Prednisone, and Rituximab in Patients With Newly Diagnosed DLBCL
Brief Title: R-CMOP in Patients With Newly Diagnosed Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024014
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-09

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Mitoxantrone hydrochloride liposome injection; Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Vincristine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-CMOP (Experimental): R-CMOP regimen includes rituximab (R), cyclophosphamide (C), mitoxantrone hydrochloride liposome injection (M), vincristine (O), and prednisone (P).
  The regimen will be administered every 3 weeks, for a maximum of 6 cycles.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome; Drug: Rituximab (R); Drug: Cyclophosphamide (CTX); Drug: Vincristin; Drug: Prednisolone

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome — assigned dose according to the 3+3 dose-escalation design in part 1, RP2D in part 2, D2
Drug: Rituximab (R) — 375mg/m2, D2
Drug: Cyclophosphamide (CTX) — 750mg/m2, D2
Drug: Vincristin — 1.2mg/m2, maximum 2mg， D2
Drug: Prednisolone — 60mg/m2, D2-6

SUMMARY:
This is a prospective clinical study to evaluate the safety and efficacy of R-CMOP in patients with newly diagnosed diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
This is an open, multicenter, prospective phase I/II clinical study to evaluate the safety and efficacy of mitoxantrone hydrochloride liposome injection in combination with cyclophosphamide, vincristine, prednisone, and rituximab (R-CMOP) in patients with newly diagnosed diffuse large B-cell lymphoma. The study is divided into two parts. The first part uses a 3+3 dose-escalation design, in which mitoxantrone hydrochloride liposome injection in the R-CMOP regimen will be administered at three different doses: 16 mg/m², 18 mg/m², and 20 mg/m², to determine the recommended Phase 2 dose (RP2D). The second part follows a single-arm design to evaluate the efficacy and safety of the R-CMOP regimen, with mitoxantrone hydrochloride liposome injection administered at the RP2D. Each cycle consists of 21 days. A maximum of 6 cycles of therapy are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Histologically confirmed newly diagnosed diffuse large B-cell lymphoma;
3. Patients must have been untreated, including chemotherapy, targeted therapy, immunotherapy, radiotherapy;
4. There must be at least one measurable lesion per the Lugano2014 criteria；
5. For lymph lesion, the long axis must be greater than 1.5cm with 18F-deoxyglucose (18FDG) PET-CT positive；
6. Ann Arbor stages II-IV；
7. ECOG score 0~2；
8. Expected survival time ≥3 months;
9. a.)Patients should meet the following requirements and must not have received treatment with cell growth factors or blood products within 14 days prior to the hematology test: Absolute value of neutrophils ≥ 1.5 × 10^9/L; Platelet ≥ 75 × 10^9/L; Hemoglobin≥80g/L. For patients with bone marrow involvement of lymphoma, the requirements are adjusted as follows: Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L; Platelet count ≥ 50 × 10^9/L; Hemoglobin level ≥ 75 g/L.

   b.)Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN; AST and ALT ≤ 5 × ULN for patients with liver involvement. Total bilirubin ≤1.5 × ULN (≤ 3 × ULN for patients with Gilbert syndrome); c.)Creatinine clearance ≥ 50 mL/min or serum creatinine ≤ 2× ULN; d.)Coagulation function: prothrombin time or activated partial thromboplastin time≤ 1.5 × ULN, and international normalized ratio ≤ 1.5;
10. Female patients of childbearing age must have a negative pregnancy test at the time of enrollment within one week. And patients must agree to use an effective method of contraception from the study initiation until at least 12 months after the last treatment;
11. Able to understand and comply with the study, and voluntarily sign informed consent; -

Exclusion Criteria:

1. Primary central nervous system DLBCL, Primary testicular large B-cell lymphoma, Primary mediastinal (thymic) large B-cell lymphoma, Lymphomatoid granulomatosis, ALK-positive large B-cell lymphoma, Plasmablastic lymphoma, HHV8-positive DLBCL, Primary effusion lymphoma, Intravascular large B-cell lymphoma, B-cell lymphoma unclassifiable between DLBCL and classical Hodgkin lymphoma, T-cell/histiocyte-rich large B-cell lymphoma, and High-grade B-cell lymphoma；
2. transformed indolent lymphoma ;
3. Patients with active central nervous system involvement;
4. History of hematopoietic stem cell transplantation;
5. Have received prior anti-lymphoma treatment, excluding short-term or low-dose corticosteroids.;
6. Used any NMPA-approved anticancer herbal medicines or proprietary Chinese medicines within 14 days prior to the first dose;
7. History of allergy and contraindications to the same class and excipients of the experimental drug;
8. Participating in any other intervention clinical trials within 4 weeks prior to the first dose except for participation in an observational (non-interventional) clinical study or the follow-up phase of an interventional study;
9. Active bacterial or viral infections requiring systemic or intravenous drug treatment.
10. History of immunodeficiency, including anti-HIV positive;
11. Active hepatitis B and C infection (defined as hepatitis B virus surface antigen positive and hepatitis B virus DNA higher than the Upper limit of normal(ULN); Hepatitis C virus antibody positive and hepatitis C virus RNA higher than the Upper limit of normal);
12. syphilis infection;
13. Individuals with an underlying medical condition, alcohol or drug abuse or dependence that impedes study drug administration or interferes with interpretation of study drug toxicity and AE, or results in inadequate or reduced adherence to the study;
14. Patients with interstitial lung disease that requires treatment; 15: A history of severe cardiovascular disease, including but not limited to:

    1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, or second to third-degree atrioventricular (AV) block;
    2. A mean QTcF interval longer than 450 ms, based on three 12-lead ECGs taken at rest;
    3. Acute coronary syndrome, congestive heart failure, stroke, or any other Grade 3 or higher cardiovascular event occurring within 6 months prior to the first dose of therapy;
    4. NYHA functional class ≥ II or left ventricular ejection fraction (LVEF)lower than 50%;
    5. Any factors that increase the risk of QTc prolongation or arrhythmias, such as heart failure, hypokalemia, congenital long QT syndrome, a family history of long QT syndrome or unexplained sudden death in a first-degree relative under the age of 40, or concurrent use of any medications known to prolong the QT interval;
    6. uncontrolled hypertension;

16. History of other malignant tumor within 2 years, except for DLBCL in this trial or resected locally cancer that has been cured (e.g.basal cell or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast); 17. No psychological, spiritual potentially hampering compliance with the study protocol and follow-up schedule; 18. Women who are pregnant or breastfeeding; 19. Any other reasons deemed by the investigator to render the participant unsuitable for inclusion in this clinical trial.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Phase I:Maximum tolerated dose (MTD) | Through the last patient complete his DLT observation, assessed up to 21 days
  Maximum tolerated dose (MTD) of liposomal mitoxantrone hydrochloride in R-CMOP
Phase I: Recommended phaseII dose (RP2D) | Through the last patient complete his DLT observation, assessed up to 21 days
  The Recommended Phase II Dose (RP2D) is defined as the optimal dose of liposomal mitoxantrone hydrochloride for use in Phase II trials, as determined by the outcomes of the Phase I study.
Phase II:Complete remission rate (CRR) | up to 2 years
  Response is assessed according to the lugano criteria
Phase I: Dose limited toxicities (DLTs) | Through the last patient complete his DLT observation, assessed up to 21 days
  adverse events defined as DLT events per protocol

SECONDARY OUTCOMES:
Phase I: The incidence rates of adverse events (AEs) | up to 2 years
  AE or severe adverse events (SAE) occur since the first dose of therapy is given
Phase I: Objective response rate (ORR) | up to 2 years
  Response is assessed according to the lugano criteria
Phase I: Complete remission rate (CRR) | up to 2 years
  Response is assessed according to the lugano criteria
Phase II: Overall response rate (ORR) | up to 2 years
  Response is assessed according to the lugano criteria
Phase II: Partial response rate (PRR) | up to 2 years
  Response is assessed according to the lugano criteria
Phase II: Duration of response (DOR) | up to 2 years
  DOR was defined as the time from first complete response or partial response to disease progression or death from any causes.
Phase II: Progression-free survival (PFS) | up to 2 years
  From the date of the first dose of therapy is given until disease progression or death from any cause.
Phase II: Overall survival (OS) | up to 2 years
  From the date of inclusion to date of death, irrespective of cause
Phase II: Disease-free survival (DFS) | up to 2 years
  From the date of achieving a complete response until disease progression or death from any cause.
Phase II: Event-free survival (EFS) | up to 2 years
  From the date of the first dose of therapy is given until disease progression, death , or the initiation of a new treatment regimen.
Phase II: The incidence rates of adverse events (AEs) | up to 2 years
  AE or severe adverse events (SAE) occur since the first dose of therapy is given

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Professor, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided